CLINICAL TRIAL: NCT00773318
Title: SPECT-CT Guided Lymphatic Mapping and Sentinel Lymphadenectomy (LM/SL) in Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 1 patient has been enrolled. No complications reported. The research team decided to terminate the clinical trial due to insufficient patients' accrual.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: London Regional Cancer Program, Canada (Other); University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Irina Rachinsky, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R-06-433; 12638 (Other: REB)
Record Dates: First submitted 2008-07-25; First posted 2008-10-16 (Estimated); Last update posted 2012-03-05 (Estimated); Status verified 2012-03

CONDITIONS: Prostate Cancer
Keywords: LM/SL; SPECT/low-dose multislice CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Patients with histologically proven AJCC stages I - II - III prostate cancer including men with clinical T3N0M0 disease, men with PSA > 10 mg/ml, and men with Gleason score of 8-10. Prostate cancer patients scheduled for prostatectomy and pelvic lymph node dissection (CLND).
  Arm A = SPECT/CT guided LM/SL versus CLND
  Interventions: Procedure: SPECT/CT guided LM/SL

INTERVENTIONS:
Procedure: SPECT/CT guided LM/SL — Detection, localization, and removal of sentinel lymph node (s) from prostate cancer guided by an integrated SPECT/low-dose multislice CT
  Other Names: Sentinel lymph node detection

SUMMARY:
Nodal staging is a key-step in pre-treatment assessment of prostate cancer. In patients with a low probability of nodal metastasis, bilateral pelvic lymphadenectomy is controversial. The large majority of them (> 80%) are free of nodal disease in obturator and external iliac stations. On the other hand, skip metastases located outside the standard lymphadenectomy may be missed, particularly in more proximal nodal stations (i.e. common iliac nodes and pre-sacral nodes).

In prostate cancer, growing data indicate the potential utility of LM/SL, particularly in patients with a low pre-test probability of nodal disease. However, very few data have been reported on the feasibility and the utility of SPECT/CT following LM/SL. In a pilot study including 11 patients with prostate cancer, Kizu and colleagues used a software image fusion from separate SPECT and CT studies. These authors concluded to the utility of image fusion to localize anatomically the SLNs. They also suggested the use of hardware fusion from a single gantry SPECT/CT device for accurate detection of SLNs. Accordingly, Corvin and colleagues recently reported the suitability of sentinel node detection in a series of 28 patients with prostate cancer; in this study, an integrated single slice SPECT/CT device was used to localize the SLNs.

In the light of the encouraging data from literature and our own preliminary clinical experience, we hypothesized that the use of integrated SPECT/low-dose multislice CT guided LM/SL may be of clinical interest in patients with prostate cancer.

DETAILED DESCRIPTION:
A multidisciplinary team (urologist, oncologist, radiologist, pathologist, and nuclear medicine) will assess the technical feasibility of LM/SL with SPECT/CT as well as its clinical potential for the staging of regional lymph nodes in 30 consecutive patients with AJCC stages I-II-III prostate cancer scheduled for prostatectomy and pelvic lymph node dissection according to the standards of care.

This is a 2-day protocol with a single isotopic tracer (Tc99m-cysteine rhenium colloids, 10-15 nm). The tracer injections will be performed under trans-rectal ultra-sound guidance (1 inj/lobe, 74MBq, 0.2 cc).

The first day or injection day (D0), an early imaging session with planar acquisitions (anterior and posterior views) will be performed within 30 min post-tracer injection. A delayed imaging session with planar and SPECT/CT acquisitions will be also performed 1 to 3 hours after tracer injection. The SPECT/CT device to be used in this research protocol is the Infinia Hawkeye 4-slice from GE Healthcare. This hybrid camera incorporates a low-dose CT with a 2.5 mA current (eff.dose < 2mSv) on a dual-head gamma camera. SPECT/CT data will be analysed on the Xeleris 2.05v (Volumetrix for Hawkeye Oncology).

The second day (D+1 post-tracer injection), all prostate cancer patients will undergo a radical prostatectomy with complete pelvic lymph node dissection (CLND). Sentinel lymph nodes (SLNs) will be detected intra-operatively by using a gamma probe (Navigator, Tyco Healthcare). In this single tracer study, SLNs are defined as hot nodes only including the hottest node and any hot node ≥ 10% of the hottest node. In this SPECT/CT protocol, additional non-radioactive nodes eventually detected on the CT component and suspicious of tumor involvement (lymphadenopathies > 1cm) will be also removed, especially lymph nodes located in unpredictable lymphatic basins. Surgery will be performed by the same surgeons.

SLNs and non-SLNs will be analyzed by the same pathologist. For SLNs, a Hematoxylin & Eosin staining (H-E) will be firstly performed. If negative, 3 more H-E stains levels will be performed and immuno-peroxidase stains for Cytokeratins AE1/AE3, PSA, and PAP. Non-SLNs will be analyzed according to the routine protocol with 3 H-E stained levels only. The SLN features will be noted: number, anatomical localization in vivo, counting rates ex vivo. The pathological characteristics of metastatic SLNs and non-SLNs will be precisely recorded: size, involvement (micro-metastases ≤ 2mm; macro-metastases; isolated tumor cells), % of nodes involved (small < 25%; moderate = 25-75%; massive > 75%).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven prostate cancer
* Initial staging (Bone scan, CT, or MRI) according to the NCCN guidelines
* Patients with AJCC stages I - II - III prostate cancer including men with clinical T3N0M0 disease, men with PSA > 10 mg/ml, and men with Gleason score of 8-10 (high grade disease)
* Prostate cancer patients will be scheduled for prostatectomy and pelvic lymph node dissection
* Informed consent signed by the patient

Exclusion Criteria:

* Patients with no histological evidence of prostate cancer
* Patient with regionally advanced disease or metastatic disease (T4, and/or N1, and/or M1)
* Patients with clinically and/or radiologically evident regional lymph node metastases
* Patients who are not scheduled for radical prostatectomy and pelvic lymph node dissection
* Patients with physical and/or psychological contraindications
* Recent studies in Nuclear Medicine with long half-time isotopes (i.e. T ½ > 48h; 111In, 67Ga, 201Tl, 131I) performed within 1 week preceding the LM/SL

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Technical feasibility and clinical utility of LM/SL with SPECT/CT in patients with early stage prostate cancer versus CLND. | 1 year - 2 years

SECONDARY OUTCOMES:
Tolerability, operating time, and complications rate of SPECT/CT guided LM/SL | 1 year - 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Irina Rachinsky, MD, MSc, Principal Investigator — The University of Western Ontario- Nuclear Medicine; Albert Driedger, MD, PhD, Study Chair — The University of Western Ontario - Nuclear Medicine; Joseph Chin, MD, PhD, Study Director — The University of Western Ontario- Urology; Madeleine Moussa, MD, Study Director — The University of Western Ontario - Pathology
Locations (1):
- University Hospital - Dpt. of Nuclear Medicine, London, Ontario, Canada

REFERENCES:
- [Background] Weckermann D, Dorn R, Trefz M, Wagner T, Wawroschek F, Harzmann R. Sentinel lymph node dissection for prostate cancer: experience with more than 1,000 patients. J Urol. 2007 Mar;177(3):916-20. doi: 10.1016/j.juro.2006.10.074. PMID 17296375
- [Background] Corvin S, Schilling D, Eichhorn K, Hundt I, Hennenlotter J, Anastasiadis AG, Kuczyk M, Bares R, Stenzl A. Laparoscopic sentinel lymph node dissection--a novel technique for the staging of prostate cancer. Eur Urol. 2006 Feb;49(2):280-5. doi: 10.1016/j.eururo.2005.08.021. Epub 2005 Dec 9. PMID 16364536
- [Background] Kizu H, Takayama T, Fukuda M, Egawa M, Tsushima H, Yamada M, Ichiyanagi K, Yokoyama K, Onoguchi M, Tonami N. Fusion of SPECT and multidetector CT images for accurate localization of pelvic sentinel lymph nodes in prostate cancer patients. J Nucl Med Technol. 2005 Jun;33(2):78-82. PMID 15930020
- [Background] Schumacher MC, Burkhard FC, Thalmann GN, Fleischmann A, Studer UE. Is pelvic lymph node dissection necessary in patients with a serum PSA<10ng/ml undergoing radical prostatectomy for prostate cancer? Eur Urol. 2006 Aug;50(2):272-9. doi: 10.1016/j.eururo.2006.01.061. Epub 2006 Feb 28. PMID 16632187
- [Background] Weckermann D, Goppelt M, Dorn R, Wawroschek F, Harzmann R. Incidence of positive pelvic lymph nodes in patients with prostate cancer, a prostate-specific antigen (PSA) level of < or =10 ng/mL and biopsy Gleason score of < or =6, and their influence on PSA progression-free survival after radical prostatectomy. BJU Int. 2006 Jun;97(6):1173-8. doi: 10.1111/j.1464-410X.2006.06166.x. PMID 16686707
- [Background] Scardino P. Update: NCCN prostate cancer Clinical Practice Guidelines. J Natl Compr Canc Netw. 2005 Nov;3 Suppl 1:S29-33. No abstract available. PMID 16280109
- [Background] de Bonilla-Damia A, Roberto Brouwer O, Meinhardt W, Valdes-Olmos RA. Lymphatic drainage in prostate carcinoma assessed by lymphoscintigraphy and SPECT/CT: its importance for the sentinel node procedure. Rev Esp Med Nucl Imagen Mol. 2012 Mar-Apr;31(2):66-70. doi: 10.1016/j.remn.2011.09.003. Epub 2011 Nov 3. PMID 22055110
- [Background] Vermeeren L, Valdes Olmos RA, Meinhardt W, Bex A, van der Poel HG, Vogel WV, Sivro F, Hoefnagel CA, Horenblas S. Value of SPECT/CT for detection and anatomic localization of sentinel lymph nodes before laparoscopic sentinel node lymphadenectomy in prostate carcinoma. J Nucl Med. 2009 Jun;50(6):865-70. doi: 10.2967/jnumed.108.060673. Epub 2009 May 14. PMID 19443579
- [Background] Krengli M, Ballare A, Cannillo B, Rudoni M, Kocjancic E, Loi G, Brambilla M, Inglese E, Frea B. Potential advantage of studying the lymphatic drainage by sentinel node technique and SPECT-CT image fusion for pelvic irradiation of prostate cancer. Int J Radiat Oncol Biol Phys. 2006 Nov 15;66(4):1100-4. doi: 10.1016/j.ijrobp.2006.06.047. Epub 2006 Sep 11. PMID 16965862
- [Background] Rousseau C, Rousseau T, Bridji B, Pallardy A, Lacoste J, Campion L, Testard A, Aillet G, Mouaden A, Curtet C, Kraeber-Bodere F. Laparoscopic sentinel lymph node (SLN) versus extensive pelvic dissection for clinically localized prostate carcinoma. Eur J Nucl Med Mol Imaging. 2012 Feb;39(2):291-9. doi: 10.1007/s00259-011-1975-x. Epub 2011 Nov 16. PMID 22086144
- See also: The University of Western Ontario — http://www.uwo.edu